CLINICAL TRIAL: NCT06637917
Title: Pulse Oximetry Performance Comparison in Newborns
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT24005PROLD
Record Dates: First submitted 2024-08-23; First posted 2024-10-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Newborn; Birth, Preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Newborn: A variety of subjects will be targeted for inclusion representing differing stages of development and environments
  Interventions: Device: OxySoftN™ Neonatal-Adult SpO2 Sensor with N600X Nellcor™ Patient Monitoring System; Device: LNCS® NEO SpO2 Sensor with RAD-97™ Pulse CO-Oximeter; Device: 1041PTS (or similar) Kendall™ Neonatal Electrodes with IntelliVue MP5 Portable Patient Monitor

INTERVENTIONS:
Device: OxySoftN™ Neonatal-Adult SpO2 Sensor with N600X Nellcor™ Patient Monitoring System — The Nellcor™ N-600x Pulse Oximetry System with N-600X Pulse Oximeter and Nellcor™ Sensors and Cables with OxiMax technology is indicated for prescription use only for the continuous non-invasive monitoring of functional oxygen saturation of arterial hemoglobin and PR. The N-600x Pulse Oximeter is intended for use with neonatal, pediatric, and adult patients during both no motion and motion conditions and for patients who are either well or poorly perfused, in hospitals, hospital-type facilities, intra-hospital transport, and home environments.
Device: LNCS® NEO SpO2 Sensor with RAD-97™ Pulse CO-Oximeter — The Masimo Rad-97™ and accessories are indicated for the continuous non-invasive monitoring of functional oxygen saturation of arterial hemoglobin, PR, carboxyhemoglobin saturation (SpCO), methemoglobin saturation (SpMet), total hemoglobin concentration (SpHb), and/or acoustic respiratory rate (RRa). The Masimo Rad-97™ and accessories are indicated for use with adult, pediatric, and neonatal patients during both no motion and motion conditions, and for patients who are well or poorly perfused. In addition, the Masimo Rad-97™ and accessories are indicated to provide the continuous non-invasive monitoring data obtained from the Masimo Rad-97™ and accessories for functional oxygen saturation of arterial hemoglobin and PR to multi-parameter devices for the display on those devices.
Device: 1041PTS (or similar) Kendall™ Neonatal Electrodes with IntelliVue MP5 Portable Patient Monitor — Market-released ECG monitoring system

SUMMARY:
The overall purpose is to directly compare pulse rate (PR) acquisition and oxygen saturation performance between two pulse oximeters (PO) in newborns.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian is willing and able to provide informed consent prior to any study procedures being performed.
* Subject is expected to be able to participate for the duration of the evaluation in the delivery room. In most instances, the length of the study will not exceed the anticipated duration of ECG monitoring.
* Subject is ≥ 29 weeks gestational age.
* Subject can accommodate multiple sensors.

Exclusion Criteria:

* Subjects that have an existing health condition, in which the investigator determines that safe or accurate oximetry measures may not be obtained at the areas where the PO sensor could be placed. For example, major congenital anomalies, limb anomalies or anyone with abrasions or surface lesions on the contact areas would be excluded.
* Any subject whose treatment or condition would be compromised if they were to participate in this study and any patient whose use of a pulse oximeter and sensor would present a potential for serious risk to health, safety, or welfare.
* Currently participating in any other study expected to confound study results in the opinion of the investigator.

Min Age: 29 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 120 newborns will be selected for this study. A variety of subjects will be targeted for inclusion representing differing stages of development and environments
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To compare time to stable signal of heart rate (HR) estimation between two pulse oximeters (PO). | Subject participation is expected to last a minimum of 5 minutes and a maximum of 12 hours.
To compare overall accuracy of heart rate (HR) estimation between two pulse oximeters (PO) as compared to gold standard electrocardiography (ECG). | Subject participation is expected to last a minimum of 5 minutes and a maximum of 12 hours.

SECONDARY OUTCOMES:
To evaluate instances of false bradycardia. | Subject participation is expected to last a minimum of 5 minutes and a maximum of 12 hours.
To evaluate instances of false bradycardia requiring emergency medical treatment. | Subject participation is expected to last a minimum of 5 minutes and a maximum of 12 hours.
To evaluate variability in PR between the two PO sensors | Subject participation is expected to last a minimum of 5 minutes and a maximum of 12 hours.
To compare the number of repositions and replacements required for the two PO sensors during monitoring. | Subject participation is expected to last a minimum of 5 minutes and a maximum of 12 hours.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cedars-Sinai, Los Angeles, California
  - Washington University in St. Louis, St Louis, Missouri
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No